CLINICAL TRIAL: NCT00891618
Title: Acupuncture for Chemo-induced Peripheral Neuropathy in Multiple Myeloma and Lymphoma Patients
Brief Title: Acupuncture for Chemo-Induced Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0679
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Lymphoma; Myeloma; Peripheral Neuropathy
Keywords: Lymphoma; Myeloma; Multiple Myeloma; MM; Non-Hodgkin's Lymphoma; NHL; Acupuncture; Treatment-induced Peripheral Neuropathy; Thalidomide; Bortezomib; Neuropathy; Peripheral Neuropathy
MeSH Terms: conditions — Lymphoma; Neoplasms, Plasma Cell; Peripheral Nervous System Diseases; Multiple Myeloma; Lymphoma, Non-Hodgkin | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acupuncture (Experimental): 3 acupuncture sessions per week for 4 weeks (Weeks 1-4), 1 week off (Week 5), then 2 per week for 4 more weeks (Weeks 6-10), total of 20 sessions. Each session lasts 20-30 minutes.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — 3 acupuncture sessions per week for 4 weeks (Weeks 1-4), 1 week off (Week 5), then 2 per week for 4 more weeks (Weeks 6-10), total of 20 sessions. Each session lasts 20-30 minutes.

SUMMARY:
The goal of this clinical research study is to learn if giving acupuncture to patients with lymphoma or a plasma cell dyscrasia can help to relieve numbness and/or tingling of the feet and/or hands that is related to chemotherapy.

DETAILED DESCRIPTION:
Acupuncture:

Acupuncture involves the insertion of small, solid, sterile needles into specific points on the skin. In this study, the needles are placed in areas that are intended to help relieve numbness and tingling of the feet and hands. Weak electrical stimulation is also applied to the needles to try to improve the treatment effects of the acupuncture.

Acupuncture Sessions:

Your first acupuncture session will be on the same day as the tests described above, if possible. (If not, it will be scheduled for another day that will be no more than about 10 days after the screening visit.)

You will have an acupuncture session 3 times per week for 4 weeks (Weeks 1-4). You will then have 1 week off (Week 5). After that, you will have an acupuncture session twice per week for 4 more weeks (Weeks 6-10). This is a total of 20 sessions. In addition to the 20 planned sessions, you may also choose to receive an optional 21st acupuncture session at the end-of-study visit that is scheduled for Week 13.

For each session, you will be placed in a comfortable position and the study doctor/acupuncturist will find points on your body where the needles will be placed. All study participants will have the needles placed at the same points on the body (the hands, feet, legs, abdomen, and scalp).

Very thin, solid, sterile, stainless steel needles will be used. All of the needles are specially made for acupuncture. The depth of the needle in the skin and the number of needles used is based on standard acupuncture procedures. The needles will remain in place for about 20-30 minutes.

Electrical stimulation will be added to some of the needles on the feet and hands. This involves placing wires on the needles, which are connected to a machine that delivers a weak electrical current through the wires. The strength of the electrical current will be changed slowly until it is at a comfortable level for you.

Study Procedures:

At each session, before you receive the acupuncture, the following procedures will be performed:

* Your vital signs will be measured.
* You will be asked about any drugs you may be taking and any side effects you may be experiencing.
* The color and coating of your tongue and the quality of your pulse will be recorded.

Once a week, you will also be asked to complete the same 3 questionnaires as you did at the beginning of the study.

Most study visits will last about 1 hour. On the weeks that you complete the questionnaires, it may add about 15-20 minutes.

During the study, you may still receive your regular pain treatments. If you are receiving Neurontin (gabapentin), Cymbalta (duloxetine), and/or Lyrica (pregabalin), you must stay on the same drug(s) until you go off this study. Minor changes in the doses of your pain treatments are allowed, but if there is a large change, you will be taken off study early.

Length of Study Participation:

You may receive up to 21 acupuncture sessions over 13 weeks. If intolerable side effects or symptoms occur, you will be taken off study early.

End-of-Study Visit:

At Week 13, or if you go off study early for any reason, you will have an end-of-study visit. If the doctor thinks it is necessary, the following procedures will be performed:

* Your medical history will be recorded.
* Your vital signs will be measured.
* You will be asked about any drugs you may be taking and any side effects you may have experienced.
* You will complete the same 3 questionnaires as before.
* The 4 nerve tests will be repeated in order to learn if there have been any changes in your nerve function.
* Your tongue and pulse will be evaluated.

After the end-of-study visit, your participation in this study will be over.

This is an investigational study. The acupuncture needles used in this study are commercially available and FDA approved. It is considered experimental, however, to use acupuncture to treat numbness and/or tingling in the feet and/or hands that is related to chemotherapy.

Up to 30 patients will take part in this study. All will be enrolled at The University of Texas (UT) MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, or the legal guardians of patients, must have the ability to understand English, sign a written informed consent document, and be willing to follow protocol requirements.
2. Age > 18 years and have a diagnosis of a plasma cell dyscrasia or lymphoma.
3. Patients must have neuropathy greater or equal to 2 according to Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0 scale in spite of previous treatment with Neurontin, Cymbalta and/or Lyrica. Patients receiving any of these drugs must remain on the same medications throughout the study period; however, minor adjustments in dosage are allowed. Patients will be removed from the study if a change in type of medication is necessary. All patients will receive treatment to both upper and lower extremities, regardless of whether or not they are experiencing symptoms in all four extremities.)
4. The patient's previous chemotherapy treatment must have included thalidomide and/or bortezomib and/or any derivatives.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
6. If the patient is a woman of child-bearing potential, she must have a negative urine pregnancy test and agree to use contraception.

Exclusion Criteria:

1. Current active treatment with thalidomide and/or bortezomib.
2. Local infection at or near the acupuncture site. (Although acupuncture is a minimally invasive procedure, patients will be excluded if there is an indication of infection.)
3. Deformities that could interfere with accurate acupuncture point location or out of energy pathway as defined by traditional acupuncture theory.
4. Concurrent use of other alternative medicines such as herbal agents, high dose vitamins and anticoagulation agents.
5. Known coagulopathy and taking heparin (including low molecular weight heparin) or Coumadin at any dose. Patients on aspirin or non-steroidal anti-inflammatories will be allowed to participate.
6. Platelets < 50 H K/UL.
7. White Blood Counts (WBCs) < 3.0 K/UL.
8. Active central nervous system (CNS) disease. (The action for acupuncture may be associated with central nervous system activity, and patients with CNS pathology may respond differently to treatment than the general population.)
9. Cardiac pacemaker.
10. Mental incapacitation or significant emotional or psychological disorder that, in the opinion of the investigators, precludes study entry. (These patients may not be able to cooperate with this slightly invasive procedure or with the data collection process.)
11. Currently pregnant or lactating females. (Certain acupuncture applications have been reported to stimulate uterine contractions and may alter lactation.)
12. Chronic alcohol use as clinically estimated by the patient's physician.
13. History of diabetic neuropathy or neuropathy related to HIV.
14. Previous acupuncture treatment for any indication within 30 days of enrollment.
15. Active treatment for lymphoma, non-Hodgkin's lymphoma or multiple myeloma.
16. Planned or actual changes in type of medications that could affect symptoms related to peripheral neuropathy (PN). Note: Minor adjustments in current medications at the time of enrollment is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wang, MD, BS, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Garcia MK, Cohen L, Guo Y, Zhou Y, You B, Chiang J, Orlowski RZ, Weber D, Shah J, Alexanian R, Thomas S, Romaguera J, Zhang L, Badillo M, Chen Y, Wei Q, Lee R, Delasalle K, Green V, Wang M. Electroacupuncture for thalidomide/bortezomib-induced peripheral neuropathy in multiple myeloma: a feasibility study. J Hematol Oncol. 2014 May 9;7:41. doi: 10.1186/1756-8722-7-41. PMID 24886772
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 30, 2009 to March 28, 2013. All recruitment done at the University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 27 participants registered, six participants were registered but excluded before treatment from the study.
Groups:
- Acupuncture: Three (3) acupuncture sessions per week for 4 weeks (Weeks 1-4), 1 week off (Week 5), then 2 per week for 4 more weeks (Weeks 6-10), total of 20 sessions. Each session lasts 20-30 minutes.
Period: Overall Study
Arm/Group | Acupuncture
Started | 21
Completed | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Acupuncture
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 64 [46 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Mean Neuropathy Severity Score (FACT-GOG-Ntx Total Score Assessment)
Description: Functional Assessment of Cancer Treatment - Gynecologic Oncology Group Neurotoxicity Scale (FACT/GOG-Ntx) Version 4 used to assess efficacy of acupuncture for treatment-induced peripheral neuropathy among multiple myeloma and/or lymphoma patients. Severity of neuropathy measured by FACT-GOG-Ntx total score assessment where 11-item questionnaire 5 point rating scale (0="not at all" and 4=equals "very much"). FACT/GOG-Ntx Total Score ranges from 0 (best possible outcome) to 44 (worst possible outcome).
Time Frame: Baseline to Week 13. Assessments at baseline, once per week during the two treatment phases of the study, and one month (week 13) after the last acupuncture treatment.
Population: Participants were excluded from primary outcome if did not complete follow up assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acupuncture
Number analyzed (Participants) | 19
units on a scale
  Baseline (n=19) | 20.8 (9.6)
  Week 4 (n=18) | 16.7 (9.4)
  Week 9 (n=15) | 9.9 (5.6)
  Week 13 (n=15) | 13.2 (8.5)

ADVERSE EVENTS:
Time Frame: Adverse Event reporting from baseline to last treatment, Week 13 of study. Total active study period was June 4, 2009 to May 09, 2011.
Arm/Group | Acupuncture
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No